CLINICAL TRIAL: NCT01388426
Title: Moisture Chamber Glasses for Dry Eye in Asian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Samanthila Waduthantri, Clinical Research Fellow, Clinical Associate, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R746
Record Dates: First submitted 2011-06-28; First posted 2011-07-06 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 7eye( Panoptx)™ Moisture chamber glasses (Experimental): 7eye( Panoptx)™
  Interventions: Device: 7eye( Panoptx)™ moisture chamber glasses

INTERVENTIONS:
Device: 7eye( Panoptx)™ moisture chamber glasses — moisture chamber glasses
  Other Names: 7eye™

SUMMARY:
Objective of this study is to evaluate the tolerance and potential benefit of moisture chamber glasses for dry eye in an Asian population. In this clinic based prospective interventional study, we aim to recruit patients (until 10 patients complete the study) who have evaporative dry eye due to exposure to environmental stress (such as frequency of out door activities) and keen to try out moisture chamber glasses/ eyewear from the dry eye clinic in Singapore National Centre. After informed consent, these patients will be prescribed 7eye( Panoptx)™ moisture chamber glasses/eyewear for 3 months and will be monitored on a diary for the amount of time wearing eyewear for 2 weeks and the number of eye drops for each type of medication used. Other outcomes will be changes in symptoms of dry eye using visual analog scale, as well as objective signs of dry eye (eg. corneal fluorescence staining and tear break up time (TBUT). As moisture chamber spectacles are currently not available as a treatment option for dry eye in Singapore, the findings of this study will give an insight to the efficacy of this new treatment modality in our population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with evaporative dry eye as assessed by the PI in the dry eye clinic and has occupational or lifestyle requirement to be exposed to a hyper-evaporative environment.

Exclusion Criteria:

1. Subjects who can't wear the eye wear as instructed in the study, or unable to complete the diary of eye wear use.
2. Subjects with eye lid or facial bone malformation
3. Subjects with a significant refractive error that warrants spectacles with a refractive power.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Percentage of time wearing moisture chamber glasses while outdoors during 2 weeks of the study. | 2 weeks during 3 months

SECONDARY OUTCOMES:
1.Number of eyedrops per day for each type of medication used at the end of study vs at the commencement of study,symptoms of dry eye (using the VAS),corneal fluorescence staining and tear break up time(TBUT). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Samanthila Waduthantri, Principal Investigator — Singapore National Eye Centre; Louis Tong, Principal Investigator — Singapore National Eye Centre; Chien Hua Tan, Study Chair — Singapore National Eye Centre
Locations (2):
- Singapore (2):
  - Singapore National Eye Center, Singapore, Singapore
  - Singapore National Eye Centre, Singapore, Singapore